CLINICAL TRIAL: NCT03494920
Title: DIRECT-SAFE: A Randomized Controlled Trial of DIRECT Endovascular Clot Retrieval Versus Standard Bridging Thrombolysis With Endovascular Clot Retrieval Within 4.5 Hours of Stroke Onset
Brief Title: DIRECT-SAFE: A Randomized Controlled Trial of DIRECT Endovascular Clot Retrieval Versus Standard Bridging Thrombolysis With Endovascular Clot Retrieval
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neuroscience Trials Australia (Other)
Collaborators: The Florey Institute of Neuroscience and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTA1601
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2021-07

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemia; Cerebral Infarction; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Pathologic Processes; Brain Infarction; Brain Ischemia; Tissue Plasminogen Activator; Plasminogen; Fibrinolytic Agents; Fibrin Modulating Agents; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia; Cerebral Infarction; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Pathologic Processes; Brain Infarction; Brain Ischemia

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to either direct endovascular clot retrieval or to bridging intravenous thrombolysis with endovascular clot retrieval.
Who Masked: Outcomes Assessor
Masking Description: Blinded core laboratory adjudications of the primary outcome. NIHSS and mRS (secondary outcomes) performed by blinded assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct endovascular clot retrieval (Other): Endovascular clot retrieval (ECR) within 4.5 hours stroke
  Interventions: Other: Direct endovascular clot retrieval
- Bridging thrombolysis followed by ECR (Other): Intravenous tPA (at the standard licensed dose of 0.9 mg/kg up to a maximum of 90mg, 10% as bolus and the remainder over 1 hour) followed by ECR
  Interventions: Other: Bridging thrombolysis followed by ECR

INTERVENTIONS:
Other: Direct endovascular clot retrieval — Direct endovascular clot retrieval within 4.5 hours of stroke onset
  Arms: Direct endovascular clot retrieval
Other: Bridging thrombolysis followed by ECR — Bridging thrombolysis followed by ECR within 4.5 hours of stroke onset
  Arms: Bridging thrombolysis followed by ECR

SUMMARY:
The study will be a multicentre, prospective, randomized, open label, blinded endpoint (PROBE) phase 3 trial (2 arm with 1:1 randomization) in ischemic stroke patients within 4.5 hours of stroke onset. Randomised patients will be stratified for site of baseline arterial occlusion into one of three groups: 1. internal carotid artery (ICA) 2. middle cerebral artery (MCA) 3. basilar artery (BA). Patients will be randomised to either bridging intravenous thrombolysis with endovascular clot retrieval (ECR), or direct endovascular clot retrieval.

DETAILED DESCRIPTION:
The DIRECT-SAFE trial will include patients with acute ischemic stroke, who are ≥18 years of age and are eligible for standard intravenous tPA therapy within 4.5 hours of stroke onset. Patients will be assessed for large vessel occlusion to determine their eligibility for randomization into the trial. Eligible vessel occlusions include the internal carotid artery, basilar artery or middle cerebral artery (M1 or M2). Patients will be consented after large vessel occlusion is confirmed based on standard care multimodal imaging.

Patients will be recruited in Australia, New Zealand, China, Taiwan, Vietnam, Singapore and Europe. Randomisation either direct to ECR or standard thrombolytic therapy and ECR shall be in a 1:1 ratio.

All patients will have a multimodal MR (or CT/CTP at investigator's discretion if MRI not possible) at 18 to 30 hours post treatment to assess reperfusion, recanalization, ischemic core growth and hemorrhagic transformation. Final follow up will occur at Day 90.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with acute ischemic stroke eligible using standard criteria to receive IV thrombolysis within 4.5 hours of stroke onset
2. Patient's age is ≥18 years
3. Intra-arterial clot retrieval treatment can commence (groin puncture) within 6 hours of stroke onset.
4. Arterial occlusion on CTA or MRA of the ICA, M1, M2 or basilar artery

Exclusion Criteria:

1. Intracranial hemorrhage (ICH) identified by CT or MRI
2. Rapidly improving symptoms at the discretion of the investigator
3. Pre-stroke mRS score of ≥ 4 (indicating previous disability)
4. Hypodensity in >1/3 MCA territory on non-contrast CT
5. Contra indication to imaging with contrast agents
6. Any terminal illness such that patient would not be expected to survive more than 1 year
7. Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.
8. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS)- ordinal analysis | 3 months
  Modified Rankin Scale (mRS) 0-2 or no change from baseline

SECONDARY OUTCOMES:
modified Rankin Scale (mRS)- ordinal analysis | 3 months
  mRS 0-1 or no change from baseline
Death | 3 months
  Death due to any cause
Angiographic reperfusion | Baseline
  Proportion of patients with good angiographic reperfusion (mTICI 2b-3)
Symptomatic intracranial haemorrhage (sICH) | 24 hours
  Proportion of patients with sICH

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mitchell, MD, Principal Investigator — Melbourne Health; Bernard Yan, MD, Principal Investigator — Melbourne Health
Locations (33):
- Australia (12):
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Mobile Stroke Unit, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- China (17):
  - Shantou Central Hospital, Shantou, Guangdong
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Wuhan Central Hospital, Wuhan, Hubei
  - The 4th Affiliated Hospital of CMU, Shenyang, Liaoning
  - Linyi People's Hospital, Linyi, Shandong
  - Shanxi People's Hospital, Shanxi, Taiyuan
  - Beijing Fengtai Youanmen Hospital, Beijing
  - Beijing Tiantin Hospital, Beijing
  - Yunfu People's Hospital, Guangdong
  - Shiyan Taihe Hospital, Hubei
  - Ningxiang People's Hospital, Hunan
  - China-Japan Union Hospital of Jilin University, Jilin
  - Maoming People's Hospital, Maoming
  - Binzhou People's Hospital, Shandong
  - Shunde Hospital of Southern Medical University, Shunde
  - Jingjiang People's Hospital, Taizhou
  - Tianjin TEDA Hospital, Tianjin
- Singapore General Hospital, Singapore, Singapore
- Vietnam (3):
  - Bach Mai Hospital, Hanoi
  - Military Hospital 103, Hanoi
  - 115 People's Hospital, Ho Chi Minh City

REFERENCES:
- [Derived] Mitchell PJ, Yan B, Churilov L, Dowling RJ, Bush SJ, Bivard A, Huo XC, Wang G, Zhang SY, Ton MD, Cordato DJ, Kleinig TJ, Ma H, Chandra RV, Brown H, Campbell BCV, Cheung AK, Steinfort B, Scroop R, Redmond K, Miteff F, Liu Y, Duc DP, Rice H, Parsons MW, Wu TY, Nguyen HT, Donnan GA, Miao ZR, Davis SM; DIRECT-SAFE Investigators. Endovascular thrombectomy versus standard bridging thrombolytic with endovascular thrombectomy within 4.5 h of stroke onset: an open-label, blinded-endpoint, randomised non-inferiority trial. Lancet. 2022 Jul 9;400(10346):116-125. doi: 10.1016/S0140-6736(22)00564-5. PMID 35810757
- [Derived] Mitchell PJ, Yan B, Churilov L, Dowling RJ, Bush S, Nguyen T, Campbell BCV, Donnan GA, Miao Z, Davis SM; DIRECT-SAFE Investigators. DIRECT-SAFE: A Randomized Controlled Trial of DIRECT Endovascular Clot Retrieval versus Standard Bridging Therapy. J Stroke. 2022 Jan;24(1):57-64. doi: 10.5853/jos.2021.03475. Epub 2022 Jan 31. PMID 35135060